CLINICAL TRIAL: NCT00323349
Title: Cues to Action in Diabetes Risk Education (CADRE): Randomized Study Assessing the Impact of Knowledge of Impaired Glucose Tolerance on Perceived Risk and Behavior Change Motivation
Brief Title: A Study of Attitudes About the Risk of Developing Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Association of Teachers of Preventive Medicine (Industry)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: TS-0931
Record Dates: First submitted 2006-05-06; First posted 2006-05-09 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Prediabetic State
Keywords: Glucose Tolerance Test; Health Knowledge, Attitudes, Practice; Motivation; Communication; Health Behavior
MeSH Terms: conditions — Prediabetic State; Behavior; Communication; Health Behavior

INTERVENTIONS:
Procedure: Oral Glucose Tolerance Testing
Behavioral: Education tailored to learning style preferences

SUMMARY:
Diabetes mellitus (DM) type 2 is well recognized as a major cause of morbidity and mortality in the United States, as well as a significant contributor to health disparities within the population. Changes in demographic and lifestyle characteristics in the population have led to a progressive increase in the prevalence of both diabetes and impaired glucose tolerance (IGT), a precursor to DM type 2. Although pharmacologic interventions have proven to be successful in blocking the progression from IGT to DM, they have not been as effective as diet and exercise modification. Studies of behavioral interventions in IGT have focused on the outcomes of improved DM risk factors and decreased progression to DM, but have either required extensive interventions that lack applicability to the general population or have utilized more modest interventions with no effect on risk factors. These studies have not included impact evaluations to assess the effect of knowledge of IGT status on motivation to change and perceived risk. This study will assess the impact of knowledge of IGT on the likelihood of altering health-related behaviors, utilizing the Health Belief Model as a conceptual framework. Subjects will be randomized to one of four treatment arms, organized in a factorial design to (1) assess the impact of OGTT testing on motivation to change behaviors and (2) evaluate the efficacy of a novel educational intervention linked to patients' learning styles. This evaluation will determine whether OGTT testing is more beneficial as a cue to action to motivate behavior change than a multifactorial assessment of diabetes risk. Additionally, the improvement in health motivation after an educational intervention is expected to be enhanced when the educational method is tailored to the individual's preferred learning style. This information will provide the foundation for more efficient behavioral interventions for patients at high risk for DM type 2.

ELIGIBILITY:
Inclusion Criteria:

* Increased risk for diabetes type 2 by one of the following characteristics: (1) BMI>30, (2) Age>45, (3) First-degree relative with type 2 diabetes, (4) History of gestational diabetes, (5) Prior elevated fasting glucose in the previous year.

Exclusion Criteria:

* History of diabetes (not gestational diabetes)
* Current laboratory results consistent with diabetes
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276
Dates: Start 2003-04; Study Completion 2004-12

PRIMARY OUTCOMES:
Scores on perceived risk scale after the intervention
Scores on motivation to change behavior scale after the intervention

SECONDARY OUTCOMES:
Scores on scales of perceived benefits of healthy lifestyle choices
Scores on scales of perceived barriers to healthy lifestyle choices

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Eizember, MD, Principal Investigator — Eastern Virginia Medical School
Locations (2):
- United States (2):
  - Ghent Family Practice, Norfolk, Virginia
  - Portsmouth Family Medicine, Portsmouth, Virginia